CLINICAL TRIAL: NCT02648165
Title: Secondary Prevention of Depression Through Group-based Acceptance and Commitment Therapy Preceded by an Experimental Attentional Bias Modification Procedure
Brief Title: Secondary Prevention of Depression Through Group-based ACT-Therapy Preceded by an Experimental ABM-Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: University of Oslo (Other); University of Oxford (Other); Karolinska Institutet (Other); Wichita State University (Other); The Hospital of Vestfold (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HSØ-2015056
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2019-04

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ABM + (Experimental): Attention Bias Modification
  Interventions: Behavioral: Attention Bias Modification
- ABM - (Sham Comparator): Sham Attention Bias Modification
  Interventions: Behavioral: Sham Attention Bias Modification
- ABM + and ACT (Experimental): Attention Bias Modification followed by Group Acceptance and Commitment Therapy
  Interventions: Behavioral: Attention Bias Modification; Behavioral: Acceptance and Commitment Therapy
- ABM - and ACT (Sham Comparator): Sham Attention Bias Modification followed by Group Acceptance and Commitment Therapy
  Interventions: Behavioral: Sham Attention Bias Modification; Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Attention Bias Modification — Computer based Attention Bias Modification
  Other Names: ABM+
  Arms: ABM +; ABM + and ACT
Behavioral: Sham Attention Bias Modification — Computer based Sham Attention Bias Modification
  Other Names: ABM-
  Arms: ABM -; ABM - and ACT
Behavioral: Acceptance and Commitment Therapy — Acceptance and Commitment Therapy delivered in a group therapy setting
  Other Names: ACT
  Arms: ABM + and ACT; ABM - and ACT

SUMMARY:
Depression (major depressive disorder; MDD) is a very common mental disorder. Research suggests that individuals with prior depressive episodes have a risk of the relapse or recurrence of MDD. Secondary prevention has been identified as a key goal in the long-term management of the disease. The current project aims to investigate whether group based Acceptance and Commitment Therapy (ACT) can reduce surrogate and clinical markers of relapse in a group highly vulnerable to depressive episodes. The group intervention will consist of eight sessions, and each group will consist of maximum 12 persons. The project also studies whether Attention Bias Modification (ABM) preceding the ACT intervention will enhance the effect. ABM will be administered over a fourteen days period prior to the ACT-intervention. Effect will be measured over a period of 12 months. The primary outcome is changes in depressive symptoms. ACT-specific secondary outcome measures are also included. Subjects with a history of major depression (n=200), currently in remission, will be recruited from Sørlandet Hospital (100 participants). Matched participants (100 participants) will be recruited at the University of Oslo. In the first phase, participants from Sørlandet hospital will be randomized to ABM treatment or control condition. In the second phase all participants from Sørlandet hospital will receive group based ACT treatment. Group based ACT and ABM represent interventions that are time and cost effective, and that could be made available to large number of individuals struggling with MDD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of major depression, currently in remission

Exclusion Criteria:

* Current or past neurological illness, bipolar disorder, psychosis or drug addiction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2015-04; Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change in residual symptoms of depression - self report | Will be measured at Baseline, immediately after ABM-intervention, then after 1 month, 2 months, 6 months, and 12 months
  Change in residual symptoms of depression as measured by Beck Depression Inventory
Change in residual symptoms of depression - clinician rating | Will be measured at Baseline, immediately after ABM-intervention, then after 1 month, 2 months, 6 months, and 12 months
  Change in residual symptoms of depression as rated by Hamilton Rating Scale for Depression

SECONDARY OUTCOMES:
Recurrence of major depressive episodes | Will be measured 12 months after baseline
  Measured by MINI structured interview
Changes in Cortisol response | Will be measured at Baseline, immediately after ABM-intervention, then after 1 month, 2 months, 6 months, and 12 months
  Cortisol measured in salvia. Samples taken in the morning on three days in succession.
Changes in symptoms of anxiety - self report | Will be measured at Baseline, immediately after ABM-intervention, then after 1 month, 2 months, 6 months, and 12 months
  Change in symptoms of anxiety as measured by Beck Anxiety Inventory
Changes in Quality of Life - self report | Will be measured at Baseline, then after 2 months, 6 months, and 12 months
  WHOQOL-BREF
Changes in Acceptance - self report | Will be measured at Baseline, then after 1 month, 2 months, 6 months, 12 months
  The 7-item Acceptance and Action Questionnaire - II (AAQ-II)
Changes in Values - self report | Will be measured at Baseline, then after 1 month, 2 months, 6 months, 12 months
  Bulls Eye
Changes in Values and committed action - self report | Will be measured at Baseline, then after 1 month, 2 months, 6 months, 12 months
  Engaged living scale
Changes in Emotional, Psychological and Social Well-Being - self report | Will be measured at Baseline, then after 1 month, 2 months, 6 months, 12 months
  Mental Health continuum - short form
Changes in Present-moment awareness and acceptance - self report | Will be measured at Baseline, then after 1 month, 2 months, 6 months, 12 months (only in ACT-arms)
  Philadelphia mindfulness scale
Changes in Cognitive fusion - self report | 1 month, 2 months, 6 months, 12 months (only in ACT-arms)
  Cognitive fusion questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Ø Haaland, PhD, Principal Investigator — Sørlandet Hospital
Locations (2):
- Norway (2):
  - Sørlandet Hospital, Department of Psychiatry, Arendal, Aust-Agder
  - University of Oslo, Department of Psychology, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ostergaard T, Lundgren T, Zettle R, Jonassen R, Harmer CJ, Stiles TC, Landro NI, Haaland VO. Acceptance and Commitment Therapy preceded by an experimental Attention Bias Modification procedure in recurrent depression: study protocol for a randomized controlled trial. Trials. 2018 Mar 27;19(1):203. doi: 10.1186/s13063-018-2515-9. PMID 29587807